CLINICAL TRIAL: NCT06567509
Title: Identification of Exercise Components of Core Stability and Their Effectiveness on Foot Posture, Foot Function, and Lower Limb Alignment in Adults With Flexible Flat Feet
Brief Title: Effectiveness of Core Stability Exercises on Foot Posture, Function and Limb Alignment in Flexible Flat Feet Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Responsible Party: Principal Investigator, Shahid Mohd Dar, Lecturer, International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IREC 2024-257
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Flexible Flatfoot
Keywords: Flexible Flatfoot; Core stability; Muscle endurance
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: This study will have two phases First phase(Pilot RCT study) Second phase (Randomized control trial)
Who Masked: Outcomes Assessor
Masking Description: In both the phases ,both groups will have different careproviders and therapists treating, so blinding is not required. But the Assessors need to be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pilot experimental group (Experimental): Phase 1: 1. Cross Curl 15 rept × 3 times 120 sec rest between the sets 2. Bridges with leg lifts 20 sec hold × 3 times 120 sec rest between the sets Side bridges (left and right) 20 sec hold × 3 times 120 sec rest between the sets 3. Planks on feet 20 sec hold × 3 times 120 sec rest between the sets 4. Quadripedal stance. 20 sec hold × 3 times 120 sec rest between the sets 5. Bicycles 15 rept × 3 times 120 sec rest between the sets
  Phase 2: 1. Cross Curl ups 20 rept × 3 times 120 sec rest between the sets 2. Bridges with leg lifts 30 sec hold × 3 times 120 sec rest between the sets Side bridges (left and right) 30 sec hold × 3 times 120 sec rest between the sets 3. Planks on feet 30 sec hold × 3 times 120 sec rest between the sets 4. Quadripedal stance 30 sec hold × 3 times 120 sec rest between the sets 5. Bicycles 20 rept × 3 times 120 sec rest between the sets
  Interventions: Other: Core stability exercises and Short foot exercises
- Pilot Control group (Other): Conventional foot exercises for control group (3 times weekly for 6 weeks)
  A. Warm up:
  Active ROM exercise (Knee and hip flexion) 10 repetitions × 2 sets)
  B. Training:
  * Active dorsiflexion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets)
  * Active plantarflexion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets)
  * Active inversion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets)
  * Active eversion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets)
  C. Cool down:
  • Calf stretches in long sitting for 10 sec hold × 3 sets.
  Interventions: Other: Conventional foot exercises and short foot exercises
- Main RCT Experimental group (Experimental): Phase 1: 1. Cross Curl 15 rept × 3 times 120 sec rest between the sets 2. Bridges with leg lifts 20 sec hold × 3 times 120 sec rest between the sets Side bridges (left and right) 20 sec hold × 3 times 120 sec rest between the sets 3. Planks on feet 20 sec hold × 3 times 120 sec rest between the sets 4. Quadripedal stance. 20 sec hold × 3 times 120 sec rest between the sets 5. Bicycles 15 rept × 3 times 120 sec rest between the sets
  Phase 2: 1. Cross Curl ups 20 rept × 3 times 120 sec rest between the sets 2. Bridges with leg lifts 30 sec hold × 3 times 120 sec rest between the sets Side bridges (left and right) 30 sec hold × 3 times 120 sec rest between the sets 3. Planks on feet 30 sec hold × 3 times 120 sec rest between the sets 4. Quadripedal stance 30 sec hold × 3 times 120 sec rest between the sets 5. Bicycles 20 rept × 3 times 120 sec rest between the sets
  Interventions: Other: Core stability exercises and Short foot exercises
- Main RCT Control Group (Other): Conventional foot exercises for control group (3 times weekly for 6 weeks)
  A. Warm up:
  Active ROM exercise (Knee and hip flexion) 10 repetitions × 2 sets)
  B. Training:
  * Active dorsiflexion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets)
  * Active plantarflexion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets)
  * Active inversion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets)
  * Active eversion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets)
  C. Cool down:
  • Calf stretches in long sitting for 10 sec hold × 3 sets.
  Interventions: Other: Conventional foot exercises and short foot exercises

INTERVENTIONS:
Other: Core stability exercises and Short foot exercises — Core stabilty exercises are the exercises where subjects will be trained to perform exercises like: Curl ups, bridging, side bridges, Planks, and Quadripedal stance exercises in a phased manner, each phase lasting 2 weeks. Complexities and duration of exercises will be increased in each phase. Short foot exercises for control group will include traditional treatment of stretching and strengthening of foot musculature.
  Arms: Main RCT Experimental group; Pilot experimental group
Other: Conventional foot exercises and short foot exercises — Ankle dorsiflexion, Plantar flexion, Inversion and Eversion range of motion exercises
  Arms: Main RCT Control Group; Pilot Control group

SUMMARY:
Flexible flat foot is a very common musculoskeletal disorder of lower limbs in general population. Studies have reported that a flexible flat foot causes an alteration in the human body structures and lower limb kinetics due to a rotational torque in the tibia and femur which in turn affects the lumbar spine. This altered mechanics affects the musculature around the lumbar spine especially the core muscles. A strong link between core muscles and lower limb control, foot posture and pressure force has been found in previous studies. While the role of core muscles on lower limb posture and functions has been determined, there is lack of evidence on the benefits of core stabilization exercises on foot arch deficits. Hence, the proposed study will determine the exercise components of core muscles training that are relevant for the flat foot pathology and then will experiment its effects on the foot posture and function. The first step of the proposed study will begin with an extensive literature survey to identify the components of core stability training that have been recommended in the management of lower limbs dysfunction. Then, a protocol of core muscles training will be devised and followed up with a pilot study where the purpose will be to assess the feasibility of the training protocol. The final step of the proposed study will be an experimental study. The subjects for the experimental study will be selected based on predetermined inclusion and exclusion criteria and will be allocated alternately into experimental and control group. The experimental group will receive core stability training as an intervention. Whereas the control group will receive traditional conventional physiotherapy treatment. The foot posture, foot function and lower limb alignment will be assessed before and after the completion of treatment protocol. The data will be analyzed for any differences between group differences and between group differences. The outcomes of the proposed study may have an implication in the lower limb alignment and foot arch correction strategies.

DETAILED DESCRIPTION:
Objective of study:

To assess effect of core stability on foot posture, function and limb alignment in adults with flexible flat feet.

Description of Methodology

The study will be conducted in the International Islamic University Malaysia (IIUM) Kuantan Campus at the research lab of the Department of Physical Rehabilitation Sciences. The pilot randomized control trial will be done to test the protocol of exercises, which were developed by authors after a systematic review. Then a randomized control trial will be conducted in the next phase.

A total of 20 Subjects with flexible flat feet will be chosen from the Kuantan community between the age group of 18 to 40 years using simple random sampling for pilot RCT and sample size for the Main RCT will be calculated after the completion of Pilot RCT.

Detailed Description of patient selection :

Subjects with flat feet will be identified from Kuantan community by one researcher using advertisement banners and inviting the general population to participate in the research and the patients will be identified using predetermined inclusion and exclusion criteria.

After that the subjects will be randomly allocated to two groups (Experimental group and control group) using random generator by one investigator, who will not be a part of assessment and administering exercises to the patients and allocation will be concealed. Then base line assessment of the patients for: Staheli Plantar arch Index, Rare foot angle, Foot function Index, Qangle, and core muscle endurance will be assessed for both the groups by an assessor who will have no role in administering exercises to the patients. Then two clinicial physiotherapists will be assigned for administering the exercises to the experimental group and control group. The clinician who will be treating the experimental group will only treat patients of the experimental group and the physiotherapist assigned to control group will be only treating patients in control group.

Details of Protocol of exercises for Pilot study:

A detailed literature survey was conducted and a systematic review was done by five researchers to identify the components of core stability exercises that may have a potential to improve lower limb function and also identify the parameters of exercise prescription. Review was conducted from December 2023 untill August 2024 and was registered with PROSPERO with registration number (CRD42023491502). Now after all the components and parameters have been identified exercises will be implemented with following details:

Pilot Experimental group:

Experimental group will undergo following components of core stability exercises : 1. Cross curl ups 2. Bridges 3. Side bridges 4. Planks 5. Quadrepedal stance 6. Bicycles.

The exercises will be implemented for a period of 6 weeks in three phases:

1. Phase 1 will last for week 1-2.
2. Phase 2 will last from week 3-4.
3. Phase 3 will last from week 5-6.

In phase 1 the exercises will be performed with 20 seconds hold for isometric contraction and 15 repetitions for isotonic component, 3 times and 120 seconds rest between the sets.

In Phase 2 same exercises will be performed with 30 seconds hold or 20 repetitions (isometric or isotonic respectively), 3 time and 120 seconds rest between the sets.

In Phase 3 same exercises will be performed with 40 seconds hold or 25 repetitions (isometric or isotonic respectively), 3 time and 120 seconds rest between the sets.

The patients will be taught the exercises in a face to face session at the start of the session and then will follow the exercises three times weekly as home exercises, i.e.... In phase 1 on Monday the patients will visit the research Lab and the assigned physiotherapist will administer the core stability exercise session and provide education about the exercise programme and then the patients will perform these exercises three time weekly for next 2 weeks. After the completion of phase 1 the patients will again visit the research Lab and assigned physiotherapist will again administer the core stability exercise session and provide education and the patients will follow the exercises three times weekly. Same procedure will be followed for the phase 3 also. For home exercises session a soft copy of pdf booklet will be circulated to the patients via a common WhatsApp group and reminders for the exercises will be given via WhatsApp group. Also a spread sheet using google forms will be created and shared with all the patients to report the attendance and to address any difficulties the subjects are facing while performing exercises in order to get the feed back about protocol.

The exercises will be preceded with a 5 minutes warm up exercises( Cat camel exercises & supine roiling) 3 times each AND end with a cool down exercise of self-stretching of hamstrings and calf in long sitting position 3 times with 10 seconds hold.

Pilot Control group:

A physiotherapist assigned for the control group will administer first session of every phase in face to face mode and the remaining sessions of the phase will be home programmed with a soft copy booklet of exercises provided to each participant via a separate WhatsApp group in a similar fashion as that of experimental group.

Pilot control group will undergo foot exercises three time weekly for a period of 6 weeks with following exercises:

Exercise session will start with arm up session of 5 minutes with Active range of motion exercises (Knee and hip flexion) 10 repetitions × 2 sets

Then a Training session for foot muscles will follow with following exercises:

Active dorsiflexion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets) Active plantarflexion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets) Active inversion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets) Active eversion exercises in long sitting (10 sec hold × 15 repetitions ×2 sets)

Finally end with Cool down of calf stretches in long sitting for 10 seconds hold × 3 sets

After the completion of six weeks of exercises, Staheli Plantar arch Index, Rare foot angle, Foot function Index, Q angle, and core muscle endurance will be again measured by the same assessor who had assessed these outcomes earlier at the baseline.

.

Details of Protocol of exercises for Main RCT:

After the completion of pilot study the feed back from the participants, which was gathered via google form will be analyzed and any fine tuning of the protocol, if required will be done and the exercises will be administered in the same fashion as mentioned in the pilot trial i.e... in nutshell two groups will be created (Experimental and control ) using random generator by one investigator and then the subjects will be assessed for the outcomes already mentioned (Staheli Plantar arch Index, Rare foot angle, Foot function Index, Q angle, and core muscle endurance) in both the groups by an assessor who will have no role in administering exercises to the patients. Then the core stability exercises and conventional foot exercises will be administered to experimental and control groups respectively by two separate physiotherapists in similar way as described in the pilot study with same parameters in three phases for 6 weeks with treatment administered three times weekly. Finally arch index, rare foot angle, foot function Index, Q angle and core muscle endurance will be again measures in both the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of age group 18 to 30 years.
2. Both males and females.
3. No recent history of lower limb injuries.
4. Subjects with bilateral flexible flat feet as per the definition.
5. Subjects with positive navicular drop test (> 10mm).
6. Subjects with Positive Jack toe rising test.

Exclusion Criteria:

1. Rigid flat foot
2. Subject who are involved in a specific sport at least 2 h /day and 3 times a week regularly.
3. History of arthritic symptoms of lower limb joints.
4. History of any ligament or tendon injuries around ankle, knee, or hip joint.
5. History of any limb surgery or back surgery.
6. Chronic back pain.
7. Any history of neurological deficit or diabetic neuropathy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Foot Posture (Staheli plantar arch index) | Will be assessed at baseline and after 6 weeks in both the groups.
  Staheli index will be calculated by a conventional footprint method. The footprints will be obtained using the standard method. Each subject will be seated and asked to stand up and press intensely over the inked rubber pad. Then will be asked to sit back to the initial position and lift their foot from the inked rubber pad. The subject will then be requested to stand steady on a plain white paper with equal pressure on both feet and then to sit again and lift his/her foot from the graph sheet. Staheli index will then be calculated as the ratio of maximal mid foot width to the maximal hind foot width. Footprint analysis using Staheli index is reported to be a valid and reliable tool.
Foot Posture (Rare foot angle) | Will be assessed at baseline and after 6 weeks in both the groups.
  The rear foot angle (RFA) will be used to assess the calcaneal valgus. Four points will be marker in the lower limb with the subject is in standing position with talus in neutral position:
  Base of calcaneus as mark 1, Subtalar joint (Centre of Achillies tendon attachment) as mark 2 and centre of posterior aspect of calf 15 cm above the 2nd mark as mark 3. A straight line will be drawn using a marker from point 2 to point 1. Then a line will be drawn from point 3 to point 2. The angle formed between the two lines with point 2 as fulcrum is the rare foot angle and will be measure using a universal goniometer.
Function (Foot function Index) | Will be assessed at baseline and after 6 weeks in both the groups.
  Foot function index questionnaire which comprises of 23 questions in the domains of pain, disability and activity limitation will be used to assess the foot function. Each question is rated from 0 (no pain or difficulty) to 10 (greatest agony) which represent the foot function in the past week. Subjects will be rated in percentage.
Lower limb alignment (Q angle) | Will be assessed at baseline and after 6 weeks in both the groups.
  The 'Q angle' will be measured by extending a line from anterior superior iliac spine of the pelvic bone to the center point of patella and extending another line from tibial tubercle of tibia to the center point of patella. The junction between these two lines is the 'Q angle' and will be measured using a universal goniometer.

SECONDARY OUTCOMES:
Core Muscle Endurance (MacGill protocol): Isometric extensor test | Will be assessed at baseline and after 6 weeks in both the groups.
  Isometric extensor test:
  The subject will lay down prone on the bed with his or her lower body from ankles to hips fixed to the testing bed. A chair of the height of the testing bed will be placed in front of the bed so that patient's upper body can be rested on. Then slowly the chair will be removed, and the patient will be asked to maintain the extension of trunk with two hands crossed over on the opposite shoulders. Time will be recorder using a stopwatch from the time the subject assumed the horizontal position till the patient deviates from the horizontal position or patient verbally quits the test.
  • Isometric flexor test: The flexor endurance will be tested by asking the subject to lay in a sit-up posture with hips and knees flexed 90 degrees and the back resting against a wedge inclined at 60 degrees and hands of subject are on the opposite shoulders with toes strapped . The posterior wedge is pulled backwards 10 cm and the subject
Core Muscle Endurance (MacGill protocol): Isometric flexor test | Will be assessed at baseline and after 6 weeks in both the groups.
  Isometric flexor test:
  The flexor endurance will be tested by asking the subject to lay in a sit-up posture with hips and knees flexed 90 degrees and the back resting against a wedge inclined at 60 degrees and hands of subject are on the opposite shoulders with toes strapped. The posterior wedge is pulled backwards 10 cm and the subject is allowed to maintain the flexed posture as long as possible and the time from the removal of wedge till any postural deviation is noted using a stop watch. Deviation is noted if the back touches the wedge.
Core Muscle Endurance (MacGill protocol): Isometric flexor test (Side bridges test, left & right) | Will be assessed at baseline and after 6 weeks in both the groups.
  Side bridges test (Left and right):
  The subject is instructed to lie inside bridge position and place one elbow 90 degrees flexed below the shoulder, and the legs are extended in line with the trunk with one foot positioned in front of the another. the second hand is crossed and kept on the opposite shoulder. The test will then be started with the patient lifting his or her pelvis from the ground and maintaining this position and the failure will be if the back no longer remains straight or if the pelvis drops to the floor. The time will be noted using a stopwatch. The test is performed for both right side and left side.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid M Dar, MPT, Principal Investigator — International Islamic University of Malaysia

REFERENCES:
- [Background] Aenumulapalli A, Kulkarni MM, Gandotra AR. Prevalence of Flexible Flat Foot in Adults: A Cross-sectional Study. J Clin Diagn Res. 2017 Jun;11(6):AC17-AC20. doi: 10.7860/JCDR/2017/26566.10059. Epub 2017 Jun 1. PMID 28764143
- [Background] Anvita Telang, & Supriya Dhumale. (2020). Comparison of Core Stability in Individuals with Flexible Flat Foot and Normal Foot. International Journal of Science and Research. 9 (5), 1232-1243.
- [Background] Brijwasi T, Borkar P. A comprehensive exercise program improves foot alignment in people with flexible flat foot: a randomised trial. J Physiother. 2023 Jan;69(1):42-46. doi: 10.1016/j.jphys.2022.11.011. Epub 2022 Dec 14. PMID 36526555
- [Background] Eloho Nyerhovwo Igbinedion, Augustina Oghenevwaerhe Jewo, God'swill Okoro, & John Chinedu Obianke. (2022). Prevalence of Flat Foot using Plantar Arch Index among Young Adults of Delta State Nigeria. Mal J Med Health Sci,18(3), 112-117.
- [Background] Khamis S, Yizhar Z. Effect of feet hyperpronation on pelvic alignment in a standing position. Gait Posture. 2007 Jan;25(1):127-34. doi: 10.1016/j.gaitpost.2006.02.005. Epub 2006 Apr 18. PMID 16621569
- [Background] Chevidikunnan MF, Al Saif A, Gaowgzeh RA, Mamdouh KA. Effectiveness of core muscle strengthening for improving pain and dynamic balance among female patients with patellofemoral pain syndrome. J Phys Ther Sci. 2016 May;28(5):1518-23. doi: 10.1589/jpts.28.1518. Epub 2016 May 31. PMID 27313363